CLINICAL TRIAL: NCT00001534
Title: Double-Blind, Placebo-Controlled Study of the Long Term Effects of Angiotensin Converting Enzyme Inhibition (Enalapril) and Angiotensin II Receptor Blockade (Losartan) on Genetically-Induced Left Ventricular Hypertrophy in Non-Obstructive HCM
Brief Title: Long Term Effects of Enalapril and Losartan on Genetic Heart Disease
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 960144; 96-H-0144
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2003-04

CONDITIONS: Hypertrophic Cardiomyopathy; Left Ventricular Hypertrophy; Myocardial Ischemia
Keywords: Genetics; Myocardial Ischemia; Diastolic Dysfunction; Renin-Angiotensin System; Hypertrophic Cardiomyopathy; Left Ventricular (LV) Hypertrophy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Hypertrophy, Left Ventricular; Myocardial Ischemia; Hypertrophy | interventions — Losartan

INTERVENTIONS:
Drug: Losartan

SUMMARY:
The human heart is divided into four chambers. One of the four chambers, the left ventricle, is the chamber mainly responsible for pumping blood out of the heart into circulation. Hypertrophic cardiomyopathy (HCM) is a genetically inherited disease causing an abnormal thickening of the heart muscle, especially the muscle making up the left ventricle. When the left ventricle becomes abnormally large it is called left ventricular hypertrophy (LVH). This condition can cause symptoms of chest pain, shortness of breath, fatigue, and heart beat palpitations.

This study is designed to compare the ability of two drugs (enalapril and losartan) to improve symptoms and heart function of patients diagnosed with hypertrophic cardiomyopathy (HCM).

Researchers have decided to compare these drugs because each one has been used to treat patients with other diseases causing thickening of the heart muscle. In these other conditions, enalapril and losartan have improved symptoms, decreased the thickness of heart muscle, improved blood flow and supply to the heart muscle, and improved the pumping action of the heart muscle.

In this study researchers will compare the effectiveness of enalapril and losartan when given separately and together to patients with hypertrophic cardiomyopathy (HCM).

DETAILED DESCRIPTION:
Hypertrophic cardiomyopathy (HCM) is a genetic cardiac disease characterized by left ventricular (LV) hypertrophy. There is often associated LV diastolic dysfunction and myocardial ischemia. The severity of the LV hypertrophy, diastolic dysfunction, and myocardial ischemia are important determinants of clinical outcomes. Angiotensin II modulates cell growth and cardiac function. There is also increasing evidence that the renin-angiotensin system (RAS) may be present in cardiac cells, and the hypertrophic action of angiotensin II could therefore be mediated by circulating or locally produced hormone. Animal and clinical studies have demonstrated that independent of their effects on systemic blood pressure, ACE inhibition and angiotensin II receptor (AT1) blockade can reduce cardiac hypertrophy, improve LV diastolic function and myocardial ischemia. AT1 blockade may be preferable to ACE inhibitors because by inhibiting angiotensin II from binding to its receptor, the system can be turned off irrespective of the source of angiotensin II. Also, there may be fewer side effects due to lack of bradykinin. This is a double-blind, placebo-controlled study that examines the abilities of enalapril (ACE inhibition) and losartan (AT1 blockade), separately or in combination, to cause regression of the cardiac hypertrophy, and to improve LV function and myocardial perfusion in non-obstructive HCM.

ELIGIBILITY:
INCLUSION CRITERIA

HCM of either gender, aged 20-55 years.

Non-dilated LV (LVIDd less than 60 mm) with LV wall thickness of greater than or equal to 16 mm measured in any LV segment by NMR.

Non-obstructive HCM: A LV outflow gradient of less than or equal to 30 mm Hg gradient at rest and less than or equal to 55 mm Hg following isoproterenol infusion to a heart rate of greater than or equal to 120 beats per minute at cardiac catheterization.

New York Heart Association functional class I-III.

Patients who have participated in the previous toxicity study may be recruited for this study, if they wish.

Patients who have previously taken an ACE inhibitor or losartan could only be included in this study, if they have been off these drugs for a period of 6 months or longer.

EXCLUSION CRITERIA

Severe cardiac symptoms at rest (NYHA IV).

LV outflow tract gradient of greater than 30 mm Hg at rest or greater than 55 mm Hg following isoproterenol infusion to a heart rate of greater than or equal to 120 beats per minute at cardiac catheterization.

Systemic diseases (respiratory, neurologic, or locomotor) that prevent exercise testing, echocardiography or NMR, MUGA, thallium studies, and cardiac catheterization.

Coronary artery disease (greater than 50% arterial luminal narrowing of a major epicardial vessel) or congenital cardiovascular abnormalities (e.g. ASD, VSD, coronary anomalies).

Chronic atrial fibrillation.

Bleeding disorder (PTT greater than 35 sec, pro time greater than 14.7 sec, platelet count less than 154 k/mm3).

Anemia (Hb less than 12.7 g/dl in males and less than 11.0 g/dl in females); renal impairment (BUN greater than 22 mg/dl and serum creatinine greater than 1.4 mg/dl); K+ less than 3.3 mmol/l or greater than 5.1 mmol/l.

Hypertension: basal systolic and diastolic pressures of greater than 160 mm Hg or greater than 95 mm Hg, respectively on two occasions separated by one hour of rest.

Hypotension: basal sitting systolic arterial pressure less than 100 mm Hg confirmed 30 minutes later.

Must have ability to estimate LV wall thickness.

Radiographic evidence of overt cardiac failure (pulmonary edema on chest X-ray).

Negative urine pregnancy test.

Pregnant or lactating female patients.

Diminished LV systolic function (resting or exercise LV ejection fractions estimated by radionuclide angiography less than 50%).

Dependence on other cardioactive drugs such as diuretics, verapamil, B-blockers, or antiarrhythmic drugs to control symptoms and arrhythmias.

Negative HIV test.

Sensitivity to ACE inhibitor e.g. angioedema.

Must have ability to set up an outpatient monitoring system.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 112
Dates: Start 1996-09; Study Completion 2003-04

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Epstein ND, Cohn GM, Cyran F, Fananapazir L. Differences in clinical expression of hypertrophic cardiomyopathy associated with two distinct mutations in the beta-myosin heavy chain gene. A 908Leu----Val mutation and a 403Arg----Gln mutation. Circulation. 1992 Aug;86(2):345-52. doi: 10.1161/01.cir.86.2.345. PMID 1638703
- [Background] Fananapazir L, Epstein ND. Genotype-phenotype correlations in hypertrophic cardiomyopathy. Insights provided by comparisons of kindreds with distinct and identical beta-myosin heavy chain gene mutations. Circulation. 1994 Jan;89(1):22-32. doi: 10.1161/01.cir.89.1.22. PMID 8281650
- [Background] Maron BJ, Bonow RO, Cannon RO 3rd, Leon MB, Epstein SE. Hypertrophic cardiomyopathy. Interrelations of clinical manifestations, pathophysiology, and therapy (1). N Engl J Med. 1987 Mar 26;316(13):780-9. doi: 10.1056/NEJM198703263161305. No abstract available. PMID 3547130